CLINICAL TRIAL: NCT04983225
Title: A Randomized, Double-blind, Blank Controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Tolerability of Initial Periodontal Therapy Combined With Human Dental Pulp Stem Cell Injection in the Treatment of Chronic Periodontitis
Brief Title: The Safety and Tolerability of Initial Periodontal Therapy Combined With Human Dental Pulp Stem Cell Injection in the Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-hDP-MSC-101
Record Dates: First submitted 2021-06-23; First posted 2021-07-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis
Keywords: Human Dental Pulp Stem Cell
MeSH Terms: conditions — Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1×10^6 cells/site group (Experimental): Human Dental Pulp Stem Cells Injection: 1×10^6 cells/periodontal defect site.
  Interventions: Drug: Human Dental Pulp Stem Cells
- 5×10^6 cells/site group (Experimental): Human Dental Pulp Stem Cells Injection: 5×10^6 cells/periodontal defect site.
  Interventions: Drug: Human Dental Pulp Stem Cells
- 1×10^7 cells/site group (Experimental): Human Dental Pulp Stem Cells Injection: 1×10^7 cells/periodontal defect site.
  Interventions: Drug: Human Dental Pulp Stem Cells
- 2×10^7 cells/two sites group (Experimental): Human Dental Pulp Stem Cells Injection: 1×10^7 cells/periodontal defect site, two locations in total, and the total cell injection volume is 2 × 10^7 cells/2 periodontal defect sites.
  Interventions: Drug: Human Dental Pulp Stem Cells
- 3~4×10^7 cells/three or four sites group (Experimental): Human Dental Pulp Stem Cells Injection: 1×10^7 cells/periodontal defect site, three or four locations in total, and the total cell injection volume is 3 × 10^7 to 4 × 10^7 cells/3 to 4 periodontal defect sites.
  Interventions: Drug: Human Dental Pulp Stem Cells
- Saline solution group (Placebo Comparator): Saline solution: 0.6mL/periodontal defect site.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Human Dental Pulp Stem Cells — Investigational drugs: based on initial periodontal therapy (supragingival cleansing, subgingival scaling and root planning), human dental pulp stem cell injection will be given for a single local injection;
  Other Names: Initial periodontal therapy
  Arms: 1×10^6 cells/site group; 1×10^7 cells/site group; 2×10^7 cells/two sites group; 3~4×10^7 cells/three or four sites group; 5×10^6 cells/site group
Other: Saline solution — Blank control: initial Basal periodontal therapy (supragingival cleansing, subgingival scaling and root planning) followed by a single local injection of normal saline.
  Other Names: Initial periodontal therapy
  Arms: Saline solution group

SUMMARY:
The principal objective of this trial is to investigate the safety and tolerability of human dental pulp stem cells injection in the treatment of chronic periodontitis. The secondary objective is to provide the basis for dosage regimen for further clinical trials and to evaluate the preliminary efficacy.

DETAILED DESCRIPTION:
Initial periodontal therapy involves cleaning, scaling and root planing. The present dose-escalating, randomized, double-blind, blank controlled clinical trial will be conducted to evaluate the safety and tolerability of dental pulp mesenchymal stem cells injection as an adjunct with Initial periodontal therapy in chronic periodontitis. Patients meeting the inclusion criteria will be assigned into five dose groups, in a 3:1 ratio within each group to treat with drug or placebo after initial periodontal therapy. The evaluation will be conducted based on safety and efficacy end points.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old (including threshold ), unlimited gender.
* Radiological examination of the periodontal defect site shows vertical bone defect, and the probing depth (PD) is 4 to 8 mm.
* Voluntarily participate in the clinical study, understand and sign the informed consent, and comply with the relevant regulations during the study period and within 18 months after the end of the study.

Exclusion Criteria:

* Subjects with severe periodontal diseases (alveolar bone resorption generally exceeds two-thirds of the tooth root length) and affects the study tooth judgment;
* The grade of studied tooth looseness ≥ grade 2 (only buccolingual movement is defined as grade 1; buccolingual and mesiodistal movement is grade 2; vertical loosening is grade 3);
* Subjects with surgical treatment of previous periodontal bone defect sites and adjacent periodontal tissues;
* Subjects with non-steroid anti-inflammatory drug, steroid hormone therapy, and/or hormone (except topical hormones) treatment, bisphosphonates within the previous 3 months before screening;
* Subjects with severe systemic infection within the previous 3 months before screening; or antibiotics treatment within 72 h before screening;
* Subjects with uncontrolled hypertension within 1 month before screening (defined as sitting systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg after receiving the optimal antihypertensive therapy);
* Subjects with systemic diseases (including but not limited to: malignant tumor or with positive tumor examination during screening, diabetes, heart failure caused by heart disease, myocardial infarction within the first 6 months before screening, angina symptoms within the first 6 months before screening, and congenital heart disease, etc.);
* Subjects who are known to be allergic to any of the materials used in the treatment;
* Subjects with the allergic constitution and previous history of allergy to blood products;
* Laboratory test (any of them meets): abnormal liver function: ALT > 80 U/L or AST > 70 U/L; abnormal renal function: serum creatinine (picric acid method) > 97 μmol/L;
* Subjects with a bleeding tendency or coagulant dysfunction (INR ≥ 1.5 × ULN, or APTT ≥ 1.5 × ULN (except the ones who are receiving anticoagulant therapy)) or serious hematologic diseases (such as grade 3 or above anemia (Hb < 80 g/L); grade 2 or above thrombocytopenia ( < 75.0 × 109 /L))
* Viral serology positive (HBsAg, HCV antibody, HIV antibody, treponema pallidum antibody) positive;
* Subjects with unprotected sex within the previous 1 month before the screening;
* Pregnant or lactating women, or subjects with a positive result of β-HCG before the screening, or subjects who are unable or unwilling to take contraceptive measures under the investigator instruction;
* Women with oral contraceptives;
* Subjects with a history of smoking addiction in the previous 12 months before the screening (the number of cigarettes smoked per day ≥ 10);
* Subjects with mental or conscious disorders;
* Subjects who participated in other clinical studies within 3 months before the screening;
* Other circumstances deemed inappropriate by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in respiration rate of Vital Signs. | within 180 days after administration.
  Respiration rate in mg(μl)/(h·g)
Changes from baseline in heart rate of Vital Signs. | within 180 days after administration.
  Heart rate in beats per minute
Changes from baseline in blood pressure of Vital Signs. | within 180 days after administration.
  Blood pressure in mmHg
Changes from baseline in body temperature of Vital Signs. | within 180 days after administration.
  Body temperature in Celsius degree
Changes from baseline in red blood cell count of Laboratory Examination | within 180 days after administration.
  Red blood cell count in whole blood is reported in the form of number.
Changes from baseline in white blood cell count of Laboratory Examination | within 180 days after administration.
  White blood cell count in whole blood is reported in the form of number.
Changes from baseline in neutrophil count of Laboratory Examination | within 180 days after administration.
  Neutrophil count in whole blood is reported in the form of number.
Changes from baseline in lymphocyte count of Laboratory Examination | within 180 days after administration.
  Lymphocyte count in whole blood is reported in the form of number.
Changes from baseline in platelet count of Laboratory Examination | within 180 days after administration.
  Platelet count in whole blood is reported in the form of number.
Changes from baseline in hemoglobin of Laboratory Examination | within 180 days after administration.
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination | within 180 days after administration.
  Prothrombin time (PT) is a screening test for exogenous coagulation factors.
Changes from baseline in INR of Laboratory Examination | within 180 days after administration.
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent.
Changes from baseline in APTT of Laboratory Examination | within 180 days after administration.
  Activated partial thromboplastin time (APTT) is a screening test for endogenous coagulation factors.
Changes from baseline in total bilirubin of Laboratory Examination | within 180 days after administration.
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in direct bilirubin of Laboratory Examination | within 180 days after administration.
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in ALT of Laboratory Examination | within 180 days after administration.
  Changes of ALT concentration (U/L) in serum will be recorded.
Changes from baseline in AST of Laboratory Examination | within 180 days after administration.
  Changes of AST concentration (U/L) in serum will be recorded.
Changes from baseline in total protein of Laboratory Examination | within 180 days after administration.
  Changes of total protein concentration (g/L) in serum will be recorded.
Changes from baseline in albumin of Laboratory Examination | within 180 days after administration.
  Changes of albumin concentration (g/L) in serum will be recorded.
Changes from baseline in total bile acid of Laboratory Examination | within 180 days after administration.
  Changes of total bile acid concentration (μmol/L) in serum will be recorded.
Changes from baseline in urea of Laboratory Examination | within 180 days after administration.
  Changes of urea concentration (mmol/L) in serum will be recorded.
Changes from baseline in creatinine of Laboratory Examination | within 180 days after administration.
  Changes of creatinine concentration (μmol/L) in serum will be recorded.
Changes from baseline in uric acid of Laboratory Examination | within 180 days after administration.
  Changes of uric acid concentration (μmol/L) in serum will be recorded.
Changes from baseline in glucose of Laboratory Examination | within 180 days after administration.
  Changes of glucose concentration (mmol/L) in serum will be recorded.
Changes from baseline in potassium of Laboratory Examination | within 180 days after administration.
  Changes of potassium concentration (mmol/L) in serum will be recorded.
Changes from baseline in sodium of Laboratory Examination | within 180 days after administration.
  Changes of sodium concentration (mmol/L) in serum will be recorded.
Changes from baseline in chlorine of Laboratory Examination | within 180 days after administration.
  Changes of chlorine concentration (mmol/L) in serum will be recorded.
Changes from baseline in CPR of Laboratory Examination | within 180 days after administration.
  C-reactive protein (CPR) is a phylogenetically highly conserved plasma protein, changes of its plasma concentration（mg/L）will be recorded.
Changes from baseline in Detection of infectious diseases of Laboratory Examination | within 180 days after administration.
  It refers to infectious diseases screening.
Changes from baseline in IgA of Laboratory Examination | within 180 days after administration.
  Changes of IgA concentration （g/L）in serum will be recorded.
Changes from baseline in IgG of Laboratory Examination | within 180 days after administration.
  Changes of IgG concentration （g/L）in serum will be recorded.
Changes from baseline in IgM of Laboratory Examination | within 180 days after administration.
  Changes of IgM concentration （g/L）in serum will be recorded.
Changes from baseline in total IgE of Laboratory Examination | within 180 days after administration.
  Changes of total IgE concentration （g/L）in serum will be recorded.
Changes from baseline in Pregnancy test of Laboratory Examination | within 180 days after administration.
  Pregnancy test will be tested in female subjects
Changes from baseline in urine specific gravity of Laboratory Examination | within 180 days after administration.
  Changes of urine specific gravity will be recorded.
Changes from baseline in urine pH of Laboratory Examination | within 180 days after administration.
  Changes of urine pH value will be recorded.
Changes from baseline in urine glucose of Laboratory Examination | within 180 days after administration.
  Changes of urine glucose will be examined by qualitative test (positive or negative).
Changes from baseline in urine protein of Laboratory Examination | within 180 days after administration.
  Changes of urine protein will be examined by qualitative test (positive or negative).
Changes from baseline in urine ketone body of Laboratory Examination | within 180 days after administration.
  Changes of urine ketone body will be examined by qualitative test (positive or negative).
Changes from baseline in urine white blood cell of Laboratory Examination | within 180 days after administration.
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative).
Changes from baseline in urine bilirubin of Laboratory Examination | within 180 days after administration.
  Changes of urine bilirubin will be examined by qualitative test (positive or negative).
Changes from baseline in urine occult blood of Laboratory Examination | within 180 days after administration.
  Changes of urine occult blood will be examined by qualitative test (positive or negative).
Changes from baseline in stool form of Laboratory Examination | within 180 days after administration.
  Stool form is classified by Bristol Stool Form Scale into 7 categories scored from 1 to 7; (1) Separate hard lumps like nuts (difficult to pass); (2) Sausage-shaped but lumpy; (3) Like a sausage but with cracks on its surface; (4) Like a sausage or snake, smooth and soft; (5) Soft blobs with clear-cut edges (passed easily); (6) Fluffy pieces with ragged edges, a mushy stool; (7) Watery, no solid pieces, entirely liquid.
Changes from baseline in stool white blood cells of Laboratory Examination | within 180 days after administration.
  White blood cell count in stools is reported in the form of number.
Changes from baseline in stool red blood cells of Laboratory Examination | within 180 days after administration.
  Red blood cell count in stools is reported in the form of number.
Changes from baseline in stool parasite egg of Laboratory Examination | within 180 days after administration.
  Parasite egg count in stools is reported in the form of number.
Changes from baseline in stool OBT of Laboratory Examination | within 180 days after administration.
  Changes of stool OBT will be examined by qualitative test (positive or negative).
Changes from baseline in ECG | within 180 days after administration.
  The cardiac rhythm is showed in ECG in the form of continuous curve. Changes of this continuous curve will be recorded.
Incidence of Treatment-Emergent Adverse Event | within 180 days after administration.
  Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events during the study period, and the severity of adverse events is determined according to the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event | within 360 days and 720 days after administration
  Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events within 360 days and 720 days after administration, and the severity of adverse events is determined according to the NCI CTCAE version 5.0.
Change from baseline in Clinical Attachment Level (AL). | at baseline, 90 days, 180 days ,360 days, 720 days.
  Clinical Attachment Level (AL) may be assessed to the nearest millimeter by means of a graduated probe and expressed as the distance in millimeters from the CEJ to the bottom of the probeable gingival/periodontal pocket.
  The clinical assessment requires the measurement of the distance from the free gingival margin (FGM) to the CEJ for each tooth surface. After this recording, AL may be calculated from the periodontal chart (i.e. PPD - distance CEJ to FGM). In cases with gingival recession, the distance FGM-CEJ turns negative and, hence, will be added to the PPD to determine AL.
Change from baseline in Probing Depth (PD). | at baseline, 90 days, 180 days ,360 days, 720 days.
  The probing depth is the distance from the gingival margin to the bottom of the gingival sulcus/pocket, is measured to the nearest millimeter by means of periodontal probe.
Change from baseline in Probing Bleeding Index （BI） | at baseline, 90 days, 180 days ,360 days, 720 days.
  A periodontal probe is inserted to the "bottom" of the gingival/periodontal pocket applying light force and is moved gently along the tooth (root) surface. If bleeding is provoked by this examination, the site examined is considered bleeding on probing-positive and, hence, inflamed. Probing Bleeding Index is divided into 5 grades: 0, 1, 2, 3 and 4.
Change from baseline in Gingival recession （GR） | at baseline, 90 days, 180 days ,360 days, 720 days.
  Exposure of the tooth through apical migration of the gingiva is called gingival recession. Recorded as the distance in millimeters from the CEJ to the gingival margin.
Change from baseline in Tooth Mobility (TM). | at baseline, 90 days, 180 days ,360 days, 720 days.
  The continuous loss of the supporting tissues during periodontal disease progression may result in increased tooth mobility, which is divided into 3 degree: I°, II°, and III°. Changes from baseline in tooth mobility will be recorded.
Changes from baseline in height of the periodontal bone defect and average density of alveolar ridge. | at baseline, 90 days, 180 days ,360 days, 720 days.
  Changes in the height of the periodontal bone defect and the mean alveolar ridge density will be detected by Cone Beam Computed Tomography (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Wang, Master, Principal Investigator — Department of Stomatology, Peking University Third Hospital, Beijing, China.
Locations (1):
- Peking University Third Hospital, Beijing, Beijng, China

IPD SHARING:
Plan to Share IPD: No